CLINICAL TRIAL: NCT07151989
Title: Influence of Original Native Mitral Valve Lesion (Stenosis or Steno-insufficiency vs. Insufficiency) on Post-implant Structural Bioprosthetic Degeneration After Mitral Valve Replacement
Acronym: DURABLE-Mitral
Status: Enrolling by invitation | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Roberto Lorusso, Prof. MD PhD, Maastricht University Medical Center
Other Study IDs: METC 2023-0324-A-1
Record Dates: First submitted 2025-03-07; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Degeneration Mitral Bioprosthesis
Keywords: Mitral bioprosthesis degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with mitral bioprosthesis replacement: All patients undergoing elective mitral valve replacement from 2012 to 2021 who met the inclusion criteria for the study (described in the dedicated section) will be enrolled in the study. These patients will be followed-up as part of routine care, and information about the clinical status, NYHA functional class, possible rehospitalization, possible cardiovascular events and postoperative echocardiography will be available for analysis. Once consent is given, and if required by local governance, pre-, intra- and post-operative data will be collected in a dedicated, structured, database.
  Interventions: Procedure: Mitral valve replacement

INTERVENTIONS:
Procedure: Mitral valve replacement — All operations were performed through median longitudinal sternotomy or mini-sternotomy.
  Intraoperative transesophageal echocardiography (TOE) was used in all patients. Arterial cannulation was central and venous cannulation was achieved with a common two-stage cannula in the right atrium. Left ventricle was vented through the right superior pulmonary vein. In minimally invasive procedures, venous cannulation was achieved percutaneously. Myocardial protection was achieved by administration of cold crystalloid or blood cardioplegia at the surgeon's discretion in an antegrade (indirect or selective) or retrograde fashion. The removal of the calcified cusps and the decalcification of the annulus was performed according to traditional techniques. All the prosthesis were be implanted with supranular technique and 2-0 U-shaped pledgeted sutures.

SUMMARY:
It aims to perform a retrospective, multi-center, observational study. All patients undergoing elective mitral valve replacement from 2012 to 2021 who met the inclusion criteria for the study (described in the dedicated section) will be enrolled in the study. These patients will be followed-up as part of routine care, and information about the clinical status, NYHA functional class, possible rehospitalization, possible cardiovascular events and postoperative echocardiography will be available for analysis. Once consent is given, and if required by local governance, pre-, intra- and post-operative data will be collected in a dedicated, structured, database.

DETAILED DESCRIPTION:
It aims to perform a retrospective, multi-center, observational study. All patients undergoing elective mitral valve replacement from 2012 to 2021 who met the inclusion criteria for the study (described in the dedicated section) will be enrolled in the study. These patients will be followed-up as part of routine care, and information about the clinical status, NYHA functional class, possible rehospitalization, possible cardiovascular events and postoperative echocardiography will be available for analysis. Once consent is given, and if required by local governance, pre-, intra- and post-operative data will be collected in a dedicated, structured, database.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients who underwent isolated mitral valve replacement for stenosis or regurgitation
* Signed informed consent, inclusive of release of medical information where required by local governance.

Exclusion Criteria:

* - Aortic and mitral valve replacement associated with surgery of ascending aorta/aortic root;
* Aortic and mitral valve replacement associated with other cardiac valve surgery (apart from arrythmia-related ablation or procedures);
* Previous cardiac surgery of any kind;
* Surgery for acute endocarditis
* Surgery for Type A aortic dissection
* Participation in another clinical trial that could interfere with the endpoints of this study.
* Pregnant or breastfeeding at time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing elective mitral valve replacement from 2012 to 2021 who met the inclusion criteria for the study (described in the dedicated section) will be enrolled in the study. These patients will be followed-up as part of routine care, and information about the clinical status, NYHA functional class, possible rehospitalization, possible cardiovascular events and postoperative 4 echocardiography will be available for analysis. Once consent is given, and if required by local governance, pre-, intra- and post-operative data will be collected in a dedicated, structured, database.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Prosthesis degeneration due to physiological deterioration | 20 years
  Echocardiographic paramters will be used.
  Quantitative and qualitative measurments swill be implied. The measurment used are listed below:
  1. Morphological Assessment (2D / 3D TTE & TEE)
     Leaflet morphology: thickness, mobility, calcification, pannus, tears, perforations.
     Bioprosthetic ring/annulus: dehiscence, rocking motion, paravalvular defects.
     Presence of thrombus, pannus, or vegetation.
     Structural valve deterioration (SVD) features: leaflet thickening, restricted opening, abnormal motion.
  2. Hemodynamic Assessment (Doppler Echocardiography)
  Mitral inflow pattern (continuous-wave Doppler across prosthesis):
  Peak velocity (m/s)
  Mean transprosthetic gradient (mmHg) - heart-rate dependent
  Pressure half-time (PHT, ms) - limited use in prosthetic valves, but can suggest stenosis
  Effective orifice area (EOA) (via continuity equation or PHT-derived, cautiously interpreted).
  Doppler Velocity Index (DVI) = LVOT VTI / Prosthetic MV VTI (helps detect obstruction independent of fl

SECONDARY OUTCOMES:
Long term survival | 20 years
  How long is the survival after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC+, Maastricht, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided